CLINICAL TRIAL: NCT01828528
Title: The Impact of Bariatric Surgery on Nonalcoholic Fatty Liver Disease and Cardiovascular Risk Utilizing Non-invasive Measures
Brief Title: Impact of Bariatric Surgery on Nonalcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-0026-ZB-CTIL
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic fatty liver disease; Nonalcoholic steatohepatitis; Obesity; Bariatric surgery; Weight loss
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Liver tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NAFLD after SG: 26 patients with NAFLD undergoing sleeve gastrectomy (SG).
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — An intra-operative liver biopsy was performed in 20 patients

SUMMARY:
The purpose of this study is to investigate the effect of weight loss rate on liver steatosis, steatohepatitis, fibrosis and cardiovascular risk at different stages before and after bariatric surgery. The investigators also aim to study the short-term effect of bariatric surgery on gastric cholecystokinin levels before and 10 days after the bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* 20≤ age ≤80
* BMI>35kg/m2
* Men and women
* Fatty infiltration in liver ultrasonography

Exclusion Criteria:

* Alcohol drinking > 140g/week
* Presence of hepatitis B or C or HIV
* Known liver disease such as:

  1. Wilson's disease
  2. hemochromatosis
  3. α1-antitrypsin deficiency
  4. autoimmune liver disease
  5. primary biliary cirrhosis
  6. primary sclerosing cholangitis)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 26 diabetic patients with NAFLD (diagnosed by ultra sound) undergoing sleeve gastrectomy (SG) at Surgery C department at Sheba Medical Center, Israel.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline liver steatosis, steatohepatitis and fibrosis at different stages after bariatric surgery, measured by non-invasive measurements as described below. | Baseline is defined as three weeks to one month before surgery. Different stages to compare to baseline are as following: 8-12 days and 12, 24 and 48 weeks after surgery.
  Measurements to be performed to assess liver disease stage at baseline and at 8-12 days and 12, 24 and 48 weeks after surgery:
  1. Blood tests of liver functions (Alanine transaminase, Aspartate transaminase, Alkaline Phosphatase, gamma-glutamyl transpeptidase, ferritin, prothrombin-time (PT), international normalized ratio (INR), Total/Direct Bilirubin, Albumin, uric acid), lipids profile (total cholesterol, triglycerides, HDL, LDL) and diabetes biomarkers (insulin, glucose, HbA1c).
  2. Blood tests of adiponectin (only at baseline and 48 weeks after surgery).
  3. Fibroscan test for quantifying liver fibrosis by means of elastography (only at baseline and 48 weeks after surgery).
  4. A blood test (FibroMax) for determining the stage and grade of liver damage (only at baseline and at 24 and 48 weeks after surgery).
  5. OWLiver® test (a serum based test that can discriminate NAFLD from steatohepatitis using metabolomics) at baseline and 48 weeks after surgery.

SECONDARY OUTCOMES:
Change of postoperative cardiovascular risk compared to baseline. | Baseline is defined as three weeks to one month before surgery. Change will be assessed 6-12 months after surgery.
  Patients will undergo brachial artery flow-mediated dilation (FMD) test (surrogate marker for endothelial function and cardiovascular risk).
Change in cholecystokinin levels before and after the surgery. | Baseline levels of cholecystokinin at 1-2 days before surgery compared to 8-12 days after surgery.
  In addition, gastric cholecystokinin levels will be measured from the removed stomach tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Ben-Ari, Prof, Principal Investigator — Director Liver Disease Center, Sheba Medical Center, Tel-Hashomer, Israel
Locations (1):
- Liver Disease Center, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel